CLINICAL TRIAL: NCT05947565
Title: Will Performing Invasive Urodynamic Study in Sitting or Standing Position Effect the Results in Males?
Brief Title: Patient Position and Invasive Urodynamic Study Results in Males
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Ersin Köseoglu, MD, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KocUrol4
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Lower Urinary Tract Symptoms; Diagnosis
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Invasive urodynamic study will be performed firstly in sitting position. Then, repeated in standing position.
  Interventions: Diagnostic Test: Invasive Urodynamic Study
- Group 2 (Active Comparator): Invasive urodynamic study will be performed firstly in standing position. Then, repeated in sitting position.
  Interventions: Diagnostic Test: Invasive Urodynamic Study

INTERVENTIONS:
Diagnostic Test: Invasive Urodynamic Study — Invasive Urodynamic Study (Filling cystometry and pressure-flow study) Under sterile conditions and at lithotomy position, an urethral and a rectal catheter will be inserted. Bladder will be filled by sterile saline slowly. The first feeling of urine, the first sensation of urination and the sensation of severe desire to urinate will be recorded step by step. Vesical, rectal and detrusor pressures will be monitorized during these period. After the strong desire to void sensation, filling cystometry phase will be completed. Sterile saline infusion is stopped.
  While the patient urinates the vesical, detrusor and rectal pressures, the maximum and average urine flow rates will be recorded.

SUMMARY:
The goal of this study is to learn whether the change or patient position might effect the results of invasive urodynamic study in males.

DETAILED DESCRIPTION:
Males will be randomised as Group 1 and Group 2. In Group 1, invasive urodynamic study will be performed first in sitting then repeated in standing position. In Group 2, invasive urodynamic study will be performed first in standing then repeated in sitting position. Results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Males over 18 years old and capable of standing during test

Exclusion Criteria:

* Patients not able to stand up during the test

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males over 18 years old and capable of standing during test
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Invasive urodynamic study | 1 day
  Sitting position
Invasive urodynamic study | 1 day
  Standing position

IPD SHARING:
Plan to Share IPD: No